CLINICAL TRIAL: NCT06314100
Title: The Effect of Aerosol Formed From Tobacco Heating Systems and Cigarette Smoking on the Microbiome of Supragingival Dental Biofilm
Brief Title: The Effect of Aerosol Formed From Tobacco Heating Systems on the Microbiome of Supragingival Dental Biofilm
Status: Completed | Type: Observational
Sponsor: University of Rijeka (Other)
Collaborators: Croatian Science Foundation (Other Government)
Responsible Party: Principal Investigator, Elvis Bozac, Teaching assistant (Department of Endodontics and Restorative dentistry), DMD, University of Rijeka
Other Study IDs: IP-2020-02-4027-EB
Record Dates: First submitted 2024-03-03; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Dental Caries
Keywords: dental caries; dental plaque; microbiota; smoking; smoking devices
MeSH Terms: conditions — Dental Caries; Dental Plaque; Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Supragingival dental biofilm samples for bacterial DNA isolation and sequencing
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- THS smokers: Each subject undergoes a routine intraoral examination and anamnesis. Samples of supragingival dental biofilm and saliva are taken for microbiological analysis
  Interventions: Device: Tobacco heating systems
- cigarette smokers: Each subject undergoes a routine intraoral examination and anamnesis. Samples of supragingival dental biofilm and saliva are taken for microbiological analysis
  Interventions: Behavioral: cigarette smoking
- nonsmokers: Each subject undergoes a routine intraoral examination and anamnesis. Samples of supragingival dental biofilm and saliva are taken for microbiological analysis
  Interventions: Behavioral: non smoking

INTERVENTIONS:
Device: Tobacco heating systems — The study aims to explore the effect of tobacco heating system consumption on microbiome of the supragingival dental biofilm and the risk of developing caries lesions
  Other Names: IQOS
  Groups: THS smokers
Behavioral: cigarette smoking — The study aims to explore the effect of cigarette smoking on microbiome of the supragingival dental biofilm and the risk of developing caries lesions
  Groups: cigarette smokers
Behavioral: non smoking — The non smoking group of subjects serve as control for the other two groups
  Groups: nonsmokers

SUMMARY:
Dental caries is a multifactorial disease primarily caused by supragingival dental biofilm. Its progression is influenced by many environmental factors, which include smoking. Tobacco heating systems (THS) are a novel tobacco product whose effect on the microbiome of the supragingival dental biofilm has not yet been investigated.

The aim of the proposed research is to determine and compare the composition of the microbiomes of the supragingival dental biofilm of THS smokers, cigarette smokers, and nonsmokers using the Next Generation Sequencing method and to assess and compare the risk of new caries lesion formation between the test groups using the Cariogram method.

The results of this research will provide insight into changes in the microbiome of the supragingival dental biofilm resulting from exposure to aerosols from tobacco combustion and tobacco heating.

DETAILED DESCRIPTION:
Dental caries is a dynamic disease caused by the presence of dental biofilm which leads to the demineralization and loss of hard dental tissues. Historically, the main microbes which were considered responsible for developing caries lesions were Streptococcus mutans and Lactobacilli, but results of recent studies have shown tha a far greater number of microorganisms and microbial interactions are present. Furthermore the progress of the disease is also affected by many environmental factors like tobacco smoking.

A wide number of studies have already confirmed a positive correlation between tobacco smoking and the incidence/presence of caries lesions in different populations of all ages. Also, invitro studies have confirmed that bacterial proliferation and metabolic activity is affected by the components, and concentrations of components of cigarette smoke, especially nicotine.

Tobacco heating systems (THS) are a relatively novel nicotine delivery product that when consumed creates an aerosol that has the same contents as cigarette smoke, but the concentration of it's components is greatly reduced. The effect of THS smoking on the bacterial microbiome of supragingival dental biofilm has not yet been researched.

In the present study a total of 60 subject have been enrolled: 20 THS smokers, 20 cigarette smokers and 20 non-smokers. Subject from each group are age and gender matched.

The goal of the study is to compare the bacterial microbiomes of supragingival dental biofilm of the 3 examined groups. This will be done by collecting supragingival dental biofilm samples, isolating bacterial DNA from them and conducting 16s RNA metagenomics through next generation sequencing.

Furthermore, caries risk assessments will be conducted through the Cariogram method . Necessary data for the Cariogram analysis is obtained through routine anamnesis, intraoral clinical examination and tests.

The results of the study will give more insight into the effects of THS and cigarette smoking on the microbiome and microbial interactions in supragingival dental biofilm.

ELIGIBILITY:
Inclusion Criteria:

* smokers of tobacco heating systems that have smoked at least 100 heating sticks during their lifetime and have smoked exclusively tobacco heating systems for at least 6 months
* cigarette smokers that have smoked at least 100 cigarettes during their lifetime and have smoked exclusively factory made cigarettes for at least 6 months
* non-smokers that have never smoked during their lifetime
* signed informed consent

Exclusion Criteria:

* use of antibiotics 3 month prior to examination and sampling
* active orthodontic treatment
* patients suffering from autoimmune diseases
* patients suffering from type II diabetes
* constant use of oral antiseptics
* use of corticosteroids of other immunosuppressive drugs/treatments
* patients who have less than 10 teeth

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In the present study a total of 60 subject are enrolled. The subjects are divided into 3 groups: tobacco heating system smokers, cigarette smokers and non-smokers. In each group there are 20 subjects which are age and gender matched.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-10-25 (Actual); Study Completion 2023-10-25 (Actual)

PRIMARY OUTCOMES:
diversity of bacterial species | baseline
  The number of different bacterial species present in the supragingival dental biofilm
abundance of bacterial species | baseline
  The quantity of each different bacterial species present in the supragingival dental biofilm
caries risk | baseline
  The risk of avoiding/developing new caries lesions calculated through the Cariogram computer application (the results are represented as chances which are expressed in percetagens(%))

CONTACTS AND LOCATIONS:
Overall Officials: Elvis Božac, DMD, Principal Investigator — Faculty of dental medicine, University of Rijeka
Locations (1):
- Faculty of dental medicine, University of Rijeka, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bozac E, Paljevic E, Sever E, Braut A, Spalj S, Persic Bukmir R. Clinical characteristics and caries risk assessment of tobacco heating systems smokers, cigarette smokers and non-smokers: a cross-sectional study. Clin Oral Investig. 2024 Jun 18;28(7):382. doi: 10.1007/s00784-024-05778-0. PMID 38888700